CLINICAL TRIAL: NCT06250803
Title: Early Versus Late Pancreatic Stent Placement for Preventing Post-ERCP Pancreatitis: a Multicentre, Randomised Trial
Brief Title: Early Pancreatic Stent Placement for Preventing PEP
Acronym: EVL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Anhui Medical University (Other)
Collaborators: The First Affiliated Hospital of Bengbu Medical University (Other); Anqing Municipal Hospital (Other); First Affiliated Hospital of Wannan Medical College (Other); Tongcheng People's Hospital of Anhui province (Unknown); Fuyang people's hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PJ 2023-14-12
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-02

CONDITIONS: Cholangiopancreatography, Endoscopic Rretrograde; Post-ERCP Pancreatitis
Keywords: Cholangiopancreatography, Endoscopic Rretrograde; pancreatic stent; post-ERCP pancreatitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: For enhanced objectivity in data analysis, the project statisticians will be blinded to the arm allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- early pancreatic stent placement (EPSP) (Experimental): a pancreatic stent will be placed immediately after endoscopic retrograde cholangiography (ERC) or endoscopic sphincterotomy (EST)
  Interventions: Device: early pancreatic stent placement (EPSP)
- late pancreatic stent placement (LPSP) (Other): a pancreatic stent will be placed after all completion of therapeutic biliary procedures, e.g. biliary stone removal or drainage
  Interventions: Device: early pancreatic stent placement (EPSP)

INTERVENTIONS:
Device: early pancreatic stent placement (EPSP) — In the EPSP group, a single pig-tail pancreatic stent (5Fr) will be inserted instantly after ERC or EST, and subsequent biliary procedures will proceed as planned. In contrast, in the LPSP group, while keeping the PD guidewire in place, a single pig-tail PD stent (5Fr) will be ultimately placed after all completion of therapeutic biliary procedures, e.g. biliary stone removal or drainage.
  Other Names: late pancreatic stent placement (EPSP)

SUMMARY:
Our aim is to compare early versus late pancreatic stent placement in preventing PEP among patients with naive papilla. The EVL trial will provide essential answers regarding the optimal timing of prophylactic pancreatic stent placement in PEP prevention.All patients with difficult biliary cannulation undergoing endoscopic retrograde cholangiopancreatography (ERCP) with pancreatic guidewire-assisted technique for biliary access will be told about the opportunity to participate in EVL research. In total, 768 patients will be randomly assigned (1:1) to two arms: (1) early pancreatic stent placement (EPSP) (a pancreatic stent will be placed immediately after endoscopic retrograde cholangiography (ERC) or endoscopic sphincterotomy (EST)) and (2) late pancreatic stent placement (LPSP) (a pancreatic stent will be placed after all completion of therapeutic biliary procedures, e.g. biliary stone removal or drainage).The primary outcome is the rate and severity of PEP. The secondary outcomes are hyperamylasemia, the rate of stenting success, and other ERCP-related adverse events (AEs).

DETAILED DESCRIPTION:
Patients with challenging biliary access using pancreatic guidewire-assisted method will be enrolled in the study. Recruitment will take place among individuals referred to the four participating centers for therapeutic biliary procedures. After obtaining signed consent forms, participants who meet all the inclusion criteria and have no exclusion criteria will be randomly grouped (with a 1:1 ratio) into EPSP and LPSP

ELIGIBILITY:
Inclusion Criteria:

Participants who fulfill all the below criteria will be enrolled: 1. with naive papilla; 2. over 18 years; 3. undergoing ERCP with pancreatic guidewire-assisted technique for biliary access; 4. providing a signed, written informed consent.

Exclusion Criteria:

Participants who meet any of the following criteria will be excluded: 1. unreachable main papillae; 2. surgically altered gastrointestinal anatomy; 3. concurrent acute pancreatitis; 4. biliary cannulation over pancreatic duct stent after precut sphincterotomy or wire-guided method (native early attribute); 5. failed biliary cannulation; 6. severe active cardiopulmonary disease; 7. breastfeeding or pregnancy; 8. ampullary tumour.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 768 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
The incidence and severity of post-ERCP pancreatitis | up to 1 months
  Patients were identified as post-ERCPpancreatitis if meeting two out of three criteria: pain consistent with acute pancreatitis; amylase or lipase>3 times normal limit; characteristic findings on imaging, in according to the Revised Atlanta International consensus.

SECONDARY OUTCOMES:
the incidence of hyperamylasemia | up to 1 months
  Asymptomatic hyperamylasemia was defined as an increase in serum amylase compared with pre-ERCP levels and beyond the upper limit of the normal range but showing no related symptoms. Serum amylase will be measured in all study patients at 3 and 24 hours after the procedure and subsequently at clinical discretion.
the rate of stenting success | Intra-procedure
the incidence of other ERCP-related adverse events | within 30 days after ERCP
  During the 30-day follow-up period,we will record other ERCP-related AEs such as gastrointestinal bleeding, cholangitis, and gastrointestinal perforation etc.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Department of Gastroenterology, The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui

IPD SHARING:
Plan to Share IPD: No
We are committed to promoting transparency and open science. Upon reasonable request and under certain conditions, individual participant data (IPD) from our study may be shared for further research. Access to the IPD will be considered on a case-by-case basis, following review and approval of a formal proposal by Qiao Mei.
  To inquire about accessing the IPD, interested parties may contact Qiao Mei at meiqiaomq@aliyun.com.
  Please note that data sharing is contingent upon meeting the criteria for ethical use, privacy, and confidentiality as outlined in our data sharing policy. Additionally, appropriate data transfer agreements may need to be established prior to sharing.

REFERENCES:
- [Result] Cotton PB, Eisen GM, Aabakken L, Baron TH, Hutter MM, Jacobson BC, Mergener K, Nemcek A Jr, Petersen BT, Petrini JL, Pike IM, Rabeneck L, Romagnuolo J, Vargo JJ. A lexicon for endoscopic adverse events: report of an ASGE workshop. Gastrointest Endosc. 2010 Mar;71(3):446-54. doi: 10.1016/j.gie.2009.10.027. No abstract available. PMID 20189503
- [Result] Yokoe M, Hata J, Takada T, Strasberg SM, Asbun HJ, Wakabayashi G, Kozaka K, Endo I, Deziel DJ, Miura F, Okamoto K, Hwang TL, Huang WS, Ker CG, Chen MF, Han HS, Yoon YS, Choi IS, Yoon DS, Noguchi Y, Shikata S, Ukai T, Higuchi R, Gabata T, Mori Y, Iwashita Y, Hibi T, Jagannath P, Jonas E, Liau KH, Dervenis C, Gouma DJ, Cherqui D, Belli G, Garden OJ, Gimenez ME, de Santibanes E, Suzuki K, Umezawa A, Supe AN, Pitt HA, Singh H, Chan ACW, Lau WY, Teoh AYB, Honda G, Sugioka A, Asai K, Gomi H, Itoi T, Kiriyama S, Yoshida M, Mayumi T, Matsumura N, Tokumura H, Kitano S, Hirata K, Inui K, Sumiyama Y, Yamamoto M. Tokyo Guidelines 2018: diagnostic criteria and severity grading of acute cholecystitis (with videos). J Hepatobiliary Pancreat Sci. 2018 Jan;25(1):41-54. doi: 10.1002/jhbp.515. Epub 2018 Jan 9. PMID 29032636
- [Result] Hakuta R, Hamada T, Nakai Y, Isayama H, Kogure H, Takahara N, Mizuno S, Yagioka H, Togawa O, Matsubara S, Ito Y, Yamamoto N, Tada M, Koike K. Early pancreatic stent placement in wire-guided biliary cannulation: A multicenter retrospective study. J Gastroenterol Hepatol. 2019 Jun;34(6):1116-1122. doi: 10.1111/jgh.14453. Epub 2018 Sep 19. PMID 30152138
- [Result] Arain MA, Freeman ML. Pharmacologic prophylaxis alone is not adequate to prevent post-ERCP pancreatitis. Am J Gastroenterol. 2014 Jun;109(6):910-2. doi: 10.1038/ajg.2014.123. PMID 24896759
- [Result] Sasahira N, Kawakami H, Isayama H, Uchino R, Nakai Y, Ito Y, Matsubara S, Ishiwatari H, Uebayashi M, Yagioka H, Togawa O, Toda N, Sakamoto N, Kato J, Koike K. Early use of double-guidewire technique to facilitate selective bile duct cannulation: the multicenter randomized controlled EDUCATION trial. Endoscopy. 2015 May;47(5):421-9. doi: 10.1055/s-0034-1391228. Epub 2015 Jan 15. PMID 25590186
- [Result] Wang P, Li ZS, Liu F, Ren X, Lu NH, Fan ZN, Huang Q, Zhang X, He LP, Sun WS, Zhao Q, Shi RH, Tian ZB, Li YQ, Li W, Zhi FC. Risk factors for ERCP-related complications: a prospective multicenter study. Am J Gastroenterol. 2009 Jan;104(1):31-40. doi: 10.1038/ajg.2008.5. PMID 19098846
- [Result] Buxbaum JL, Freeman M, Amateau SK, Chalhoub JM, Coelho-Prabhu N, Desai M, Elhanafi SE, Forbes N, Fujii-Lau LL, Kohli DR, Kwon RS, Machicado JD, Marya NB, Pawa S, Ruan WH, Sheth SG, Thiruvengadam NR, Thosani NC, Qumseya BJ; (ASGE Standards of Practice Committee Chair). American Society for Gastrointestinal Endoscopy guideline on post-ERCP pancreatitis prevention strategies: summary and recommendations. Gastrointest Endosc. 2023 Feb;97(2):153-162. doi: 10.1016/j.gie.2022.10.005. Epub 2022 Dec 12. No abstract available. PMID 36517310
- [Result] ASGE STANDARDS OF PRACTICE COMMITTEE; Buxbaum JL, Freeman M, Amateau SK, Chalhoub JM, Chowdhury A, Coelho-Prabhu N, Das R, Desai M, Elhanafi SE, Forbes N, Fujii-Lau LL, Kohli DR, Kwon RS, Machicado JD, Marya NB, Pawa S, Ruan WH, Sadik J, Sheth SG, Thiruvengadam NR, Thosani NC, Zhou S, Qumseya BJ; (ASGE Standards of Practice Committee Chair). American Society for Gastrointestinal Endoscopy guideline on post-ERCP pancreatitis prevention strategies: methodology and review of evidence. Gastrointest Endosc. 2023 Feb;97(2):163-183.e40. doi: 10.1016/j.gie.2022.09.011. Epub 2022 Dec 12. No abstract available. PMID 36517309
- [Result] Dumonceau JM, Kapral C, Aabakken L, Papanikolaou IS, Tringali A, Vanbiervliet G, Beyna T, Dinis-Ribeiro M, Hritz I, Mariani A, Paspatis G, Radaelli F, Lakhtakia S, Veitch AM, van Hooft JE. ERCP-related adverse events: European Society of Gastrointestinal Endoscopy (ESGE) Guideline. Endoscopy. 2020 Feb;52(2):127-149. doi: 10.1055/a-1075-4080. Epub 2019 Dec 20. PMID 31863440
- [Result] Easler JJ, Fogel EL. Prevention of post-ERCP pancreatitis: the search continues. Lancet Gastroenterol Hepatol. 2021 May;6(5):336-337. doi: 10.1016/S2468-1253(21)00063-7. Epub 2021 Mar 19. No abstract available. PMID 33740414
- [Result] Thiruvengadam NR, Kochman ML. Emerging Therapies to Prevent Post-ERCP Pancreatitis. Curr Gastroenterol Rep. 2020 Nov 13;22(12):59. doi: 10.1007/s11894-020-00796-w. PMID 33188441
- [Result] Luo H, Zhao L, Leung J, Zhang R, Liu Z, Wang X, Wang B, Nie Z, Lei T, Li X, Zhou W, Zhang L, Wang Q, Li M, Zhou Y, Liu Q, Sun H, Wang Z, Liang S, Guo X, Tao Q, Wu K, Pan Y, Guo X, Fan D. Routine pre-procedural rectal indometacin versus selective post-procedural rectal indometacin to prevent pancreatitis in patients undergoing endoscopic retrograde cholangiopancreatography: a multicentre, single-blinded, randomised controlled trial. Lancet. 2016 Jun 4;387(10035):2293-2301. doi: 10.1016/S0140-6736(16)30310-5. Epub 2016 Apr 28. PMID 27133971
- [Result] Elmunzer BJ, Scheiman JM, Lehman GA, Chak A, Mosler P, Higgins PD, Hayward RA, Romagnuolo J, Elta GH, Sherman S, Waljee AK, Repaka A, Atkinson MR, Cote GA, Kwon RS, McHenry L, Piraka CR, Wamsteker EJ, Watkins JL, Korsnes SJ, Schmidt SE, Turner SM, Nicholson S, Fogel EL; U.S. Cooperative for Outcomes Research in Endoscopy (USCORE). A randomized trial of rectal indomethacin to prevent post-ERCP pancreatitis. N Engl J Med. 2012 Apr 12;366(15):1414-22. doi: 10.1056/NEJMoa1111103. PMID 22494121
- [Result] Akshintala VS, Kanthasamy K, Bhullar FA, Sperna Weiland CJ, Kamal A, Kochar B, Gurakar M, Ngamruengphong S, Kumbhari V, Brewer-Gutierrez OI, Kalloo AN, Khashab MA, van Geenen EM, Singh VK. Incidence, severity, and mortality of post-ERCP pancreatitis: an updated systematic review and meta-analysis of 145 randomized controlled trials. Gastrointest Endosc. 2023 Jul;98(1):1-6.e12. doi: 10.1016/j.gie.2023.03.023. Epub 2023 Mar 31. PMID 37004815
- [Derived] Wang S, Bai B, Hong J, Xu W, Shen Z, Xue Y, Zhang Y, Li M, Huang Q, Zhang W, Jie L, Shi C, Hu C, Wang B, Ding H, Li S, Li D, Lu Q, Li Y, Liu X, Hong R, Mei Q, Bao J. Early versus late pancreatic stent placement for preventing post-ERCP pancreatitis: protocol of a multicenter randomized clinical trial. Trials. 2025 Jun 4;26(1):189. doi: 10.1186/s13063-025-08878-8. PMID 40462140